CLINICAL TRIAL: NCT01475864
Title: Prospective Evaluation of the Clinical Utility of Endoscopically-placed Self Expandable Stents
Brief Title: Prospective Evaluation of the Covered Self-expandable Metal Stents (CSEMS) for Incomplete Biliary Stone Clearance
Status: Withdrawn | Type: Observational
Why Stopped: no subjects were found who met criteria
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: Biliary stone
Record Dates: First submitted 2011-11-16; First posted 2011-11-21 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Choledocholithiasis
Keywords: Choledocholithiasis; metal stents; biliary duct stent
MeSH Terms: conditions — Choledocholithiasis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Incomplete biliary stone extraction.
  Interventions: Procedure: ERCP with metal stent

INTERVENTIONS:
Procedure: ERCP with metal stent — ERCP will be used so that a metal stent can be placed to facilitate the removal of the biliary stone
  Other Names: see above information

SUMMARY:
The current standard of care for bile duct stone are endoscopic sphincterotomy and stone extraction. Placement of plastic stents is an option for incomplete biliary stone clearance. This study will use the CSEMS in patients with complex biliary stones who failed stone extraction as they have the advantage of large stent diameter. CSEMS may offer a temporizing measure that allows more successful subsequent stone clearance. However, their use in benign condition has been limited especially for biliary stone removal. The purpose of this study is to determine the feasibility, safety, easy removability, stent-stone formation rate, and migration rate of CSEMS for complex biliary stones.

DETAILED DESCRIPTION:
same as brief summary

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Bilary stone unable to be extracted with balloon, basket, large balloon dilation of the ampulla or mechanical lithotripsy.
* Stone can be bridged by the metal stent
* Subject must be able to give informed consent.

Exclusion Criteria:

* Any contraindication to ERCP
* Patient refuses consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those patients who have a biliary stone that has not been removed by standard medical care.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
complete biliary stone clearance | 12 months
  This is an observational study where the ERCP being done is part of the standard of care for choledocholithiasis. There are no study interventions

SECONDARY OUTCOMES:
other techniques used for stone clearance | 12 months
  This will include the number of ERCP's needed to achive the complete biliary stone clearance, Use of mechanical Lithotripsy, use of cholangioscopy, procedure duration and any adverse events safety

CONTACTS AND LOCATIONS:
Overall Officials: Peter V Draganov, MD, Principal Investigator — University of Florida